CLINICAL TRIAL: NCT00431197
Title: Steady-State Feedback Actions of Testosterone on Luteinizing Hormone Secretion in Young and Older Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 344-03; Minn # 22270
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Ketoconazole

INTERVENTIONS:
Drug: Ketoconazole, Dexamethesone, Androgel,GnRH

SUMMARY:
This study is being done to learn how the male hormone , testosterone, affects pituitary hormones in younger and older men. The pituitary is a gland in the brain that secretes hormones, some of which normally control growth and fertility.

DETAILED DESCRIPTION:
Concentrations of bioavailable testosterone decline by 1.0-1.5% annually as men age. Reduced systemic testosterone availability is associated with decreased muscle mass, strength and aerobic capacity, decreased bone-mineral density and increased risk of hip fracture, waning sexual interest, inpaired spatial cognition and increased risk of visceral obesity, impaired glucose tolerance and coronary artery disease. Luteinizing hormone (LH) secretion often fails in healthy older individuals. In addition, aging is marked by an acceleration of LH pulse frequency, loss of high-amplitude LH pulses and disorderly release of LH and testosterone, as measured by the approximate entropy statistic. The mechanisms that underlie such complex adaptations are not known, but appear to involve multiple loci of regulatory failure.

ELIGIBILITY:
* Healthy Men Ages 18-80
* All ethnicities eligible
* Men with indeterminate erectile dysfunction eligible with normal serum gonadotropin, total testosterone, prolactin and TSH concentrations and documented integrity of the neurovascular, cardiovascular, hepatorenal systems

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
LH and Testosterone levels will be evaluated after 4 study visits

CONTACTS AND LOCATIONS:
Overall Officials: Johannes D. Veldhuis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic and Foundation, Rochester, Minnesota, United States